CLINICAL TRIAL: NCT07320300
Title: Evaluation of Post-Stroke Cognitive Impairment in Patients Attending the Neuropsychiatry Department- Assiut University
Brief Title: Post Stroke Cognitive Impairment
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kamal Eldin Mohamed Ali Ahmed, resident doctor, Assiut University
Other Study IDs: post stroke cognition
Record Dates: First submitted 2025-11-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cognition - Other
MeSH Terms: interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cognitive assessment: Montreal Cognitive Assessment (MoCA), Cognitive Assessment for Stroke patients, Oxford cognitive screening, Trail Making Test B, Digit Span-Backward, verbal fluency, Clinical Dem — Follow-up: for cognitive and functional reassessment

SUMMARY:
clinical evaluation of the prevalence and severity of cognitive impairment among patients after ischemic and haemorrhagic stroke admitted to the Neuropsychiatry department

ELIGIBILITY:
Inclusion Criteria:

Patients of both sexes, aged 18- 60 years, with a history of first stroke within 3 months of admission, all types of stroke confirmed by imaging (ischemia, parenchymal haemorrhage, subarachnoid haemorrhage, venous stroke)

Exclusion Criteria:

* Age above 60 years, refusal to participate in the study, pre-existing dementia or significant psychiatric illness, severe aphasia or communication deficits precluding cognitive testing or severe comorbid condition limiting follow-ups, systemic diseases that are known to affect the central nervous system, such as (thyroid dysfunction, chronic infections, or system failure like liver or renal failure), significant sensory impairment (deafness and blindness), history of malignancy and those who have had neurosurgical procedures or severe head trauma at any time before a stroke.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: egyptian population
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
the prevalence of cognitive impairment among patients after ischemic and haemorrhagic stroke admitted to the Neuropsychiatry department | baseline
  clinical evaluation of the prevalence of cognitive impairment among patients after ischemic and haemorrhagic stroke admitted to the Neuropsychiatry departmen
prevalence estimates of PSCI within the stroke population admitted to a tertiary hospital. | baseline

IPD SHARING:
Plan to Share IPD: Undecided